CLINICAL TRIAL: NCT02346604
Title: Pulmonary Gas Exchange Abnormalities in Patients With Mild COPD
Status: Completed | Type: Observational
Sponsor: Queen's University (Other)
Collaborators: Ontario Lung Association (Other)
Responsible Party: Principal Investigator, Dr. Denis O'Donnell, Principal Investigator, Queen's University
Other Study IDs: DMED-1458-12
Record Dates: First submitted 2015-01-07; First posted 2015-01-27 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: COPD
Keywords: exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mild COPD: Symptomatic smokers with mild COPD
- Healthy Control: Non-smokers, matched to mild COPD group for age (at least 50 years) and gender

SUMMARY:
People with mild chronic obstructive pulmonary disease (COPD) can have significant physiological abnormalities and breathing inefficiency which become more pronounced during the stress of exercise, leading to intolerable breathing discomfort (dyspnea). To better understand the mechanisms of respiratory symptoms and exercise limitation in mild COPD, we will examine detailed lung function tests and other important measurements during rest and exercise in people with mild COPD compared with healthy non-smokers. This will be the first study to uncover the fundamental causes of breathing inefficiency and the related shortness of breath during physical exertion in patients with mild COPD. We hope to demonstrate that one simple measurement during exercise [the relation (ratio) between the total amount of air breathed (ventilation) and the amount of carbon dioxide breathed out] gives meaningful information about the extent of damage to the small airways and blood vessels in mild COPD and the overall gas exchanging function of the lungs, without the need for an arterial blood sample.

This is a case-controlled observational study not involving an intervention. Participants will complete 2 visits approximately 1 week apart, each conducted at the same time of day. Visit 1 will consiste of screening for iligibility, symptom and activity assessments, pulmonary function tests and an incremental cycle cardiopulmonary exercise test (CPET) for familiarization purposes. Visit 2 will include spirometry followed by an incremental cycle CPET with detailed measures of ventilatory, gas exchange, sensory-perceptual and arterial blood gas responses.

ELIGIBILITY:
Inclusion Criteria:

* Stable symptomatic patients with GOLD grade 1B mild COPD;
* at least 50 years of age;
* a cigarette smoking history ≥20 pack-years;
* a Baseline Dyspnea Index focal score ≤9;
* post-bronchodilator forced expiratory volume in 1 second (FEV1) ≥80 %predicted and an FEV1/forced vital capacity (FVC) ratio <0.7 and < lower limit of normal.

Exclusion Criteria:

* clinically significant comorbidities;
* contraindications to exercise testing;
* history/clinical evidence of asthma;
* body mass index <18.5 or >30 kg/m2;
* use of supplemental oxygen.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients fitting GOLD grade 1B criteria for mild COPD
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2013-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
ventilatory equivalent for carbon dioxide (VE/VCO2) | Measured at its nadir during an exercise test. Participants will be followed for the amount of time taken to complete 2 study visits, an expected average duration between 1 and 2 weeks.
  Exercise will consist of a symptom-limited incremental test on a cycle ergometer

SECONDARY OUTCOMES:
dead space to tidal volume ratio (VD/VT) | Measured at standardized work rates during exercise
arterial blood gas measurements | Measured at standardized work rates during exercise
  Measurements will include arterial oxygen tension (PaO2), arterial carbon dioxide tension (PaCO2), pH, hydrogen ion (H+), plasma bicarbonate (HCO3-) and lactate.
dyspnea intensity measured using the modified 10-point Borg scale | Measured at standardized work rates during exercise

CONTACTS AND LOCATIONS:
Overall Officials: Denis E O'Donnell, MD, FRCPC, Principal Investigator — Queen's University and Kingston General Hospital
Locations (1):
- Respiratory Investigation Unit at Kingston General Hospital, Kingston, Ontario, Canada